CLINICAL TRIAL: NCT00754923
Title: A Phase II Study of Single Agent Sorafenib in Non-small Cell Lung Cancer Patients Who Never Smoked or Were Former Light Smokers.
Brief Title: Sorafenib in Treating Non-Smokers or Former Light Smokers With Relapsed or Refractory Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-08017; NCI-2011-03192 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment: Sorafenib (Experimental): Sorafenib will be administered at a dose of 400 mg taken twice daily, continuously on a 28 day cycle.
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sorafenib — administered orally at 400 mg taken twice daily , continuously on a 28 day cycle as an outpatient.
  Other Names: Nexavar; sorafenib tosylate

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sorafenib works in treating non-smokers or former light smokers with relapsed or refractory stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of sorafenib tosylate, in terms of 6-month progression-free survival rate, in non-smokers or former light smokers with relapsed or refractory stage IIIB or IV non-small cell lung cancer.

Secondary

* To determine the 1-year survival rate in patients treated with this drug.
* To assess the frequency and severity of adverse events associated with this drug in these patients.
* To investigate the mutational status of EGFR (epidermal growth factor receptor), ALK (anaplastic lymphoma kinase), ROS1, and K-Ras(Kirsten rat sarcoma viral oncogene homolog)in archived tumor samples from these patients.

OUTLINE: Patients receive oral sorafenib tosylate twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Archived tumor tissue samples are analyzed for mutations of EGFR, ALK, ROS1, and K-Ras by PCR (polymerase chain reaction) and DNA (deoxyribonucleic acid) sequencing.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * Stage IIIB or IV disease
  * Recurrent disease after prior surgery, chemotherapy, or radiotherapy
  * No squamous cell histology or mixed tumor with > 50% squamous cells
* Non-smoker (smoked ≤ 100 cigarettes in lifetime) OR former light smoker (smoked > 100 cigarettes but ≤ 10 pack years AND quit smoking ≥ 1 year ago)
* No known brain metastasis

  * Patients with neurological symptoms must undergo a CT scan or MRI of the brain to exclude brain metastasis

PATIENT CHARACTERISTICS:

* ECOG(Eastern Cooperative Oncology Group)performance status 0-2
* ANC (Absolute Neutrophil Count)≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* ALT (Alanine Aminotransferase Test) and AST (Aspartate Aminotransferase Test) ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 1.5 mg/dL
* Creatinine clearance ≥ 50 mL/min
* INR (International Normalized Ratio) < 1.5 OR PT/PTT (Prothrombin time/partial thromboplastin time)normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception prior to, during, and for ≥ 3 months after completion of study treatment
* No cardiac disease, including any of the following:

  * New York Heart Association class III-IV congestive heart failure
  * Unstable angina (anginal symptoms at rest)
  * New-onset angina within the past 3 months
  * Myocardial infarction within the past 6 months
* No cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* No uncontrolled hypertension (i.e., systolic blood pressure [BP] > 150 mm Hg or diastolic BP > 90 mm Hg) despite optimal medical management
* No thrombolic or embolic events (e.g., cerebrovascular accident, including transient ischemic attacks) within the past 6 months
* No pulmonary hemorrhage or bleeding event ≥ CTCAE (Common Terminology Criteria for Adverse Events)grade 2 within the past 4 weeks
* No other hemorrhage or bleeding event ≥ CTCAE grade 3 within the past 4 weeks
* No active clinically serious infection > CTCAE grade 2
* No serious non-healing wound, ulcer, or bone fracture
* No evidence or history of bleeding diathesis or coagulopathy
* No known HIV infection or chronic hepatitis B or C
* No other malignancy except for any of the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Other cancer from which the patient has been disease-free for ≥ 5 years with a low probability of recurrence
* No condition that impairs the patient's ability to swallow whole pills
* No malabsorption problems
* No known or suspected allergy to sorafenib tosylate or any agent given in the course of this study
* No significant traumatic injury within the past 4 weeks

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than one prior systemic chemotherapy treatment for metastatic disease

  * Prior treatment with EGFR inhibitors is not considered chemotherapy
* More than 4 weeks since prior major surgery or open biopsy
* No prior sorafenib tosylate
* No concurrent St. John's wort or rifampin
* Concurrent anticoagulation with warfarin or heparin allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A. Villalona, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment: Sorafenib
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment: Sorafenib
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 70 [49 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions", or similar definition as accurate and appropriate
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Treatment: Sorafenib
Number analyzed (Participants) | 11
participants | 11

2. Secondary Outcome: Overall Survival Rate
Description: Determine the one year survival rate in Non/Light smokers with advanced and previouslytreated NSCLC
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment: Sorafenib
Number analyzed (Participants) | 11
months | 8.8 [2.4 to 16.8]

3. Secondary Outcome: Incidence of Adverse Events Sssessed by Common Terminology Criteria for Adverse Events (CTCAE)
Description: Assess the frequency and severity of adverse events associated with Sorafenib in this patient population Non/Light smokers with advanced and previously treated NSCLC.
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment: Sorafenib
Number analyzed (Participants) | 11
percentage of participants
  Fatigue | 9
  Rash | 55

4. Secondary Outcome: Mutational Status for EGFR or Kras
Time Frame: up to 2 years
Measure: Number; unit: participants
Arm/Group | Treatment: Sorafenib
Number analyzed (Participants) | 7
participants | 7

ADVERSE EVENTS:
Arm/Group | Treatment: Sorafenib
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Sorafenib (N=11)
Fatigue (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: Sorafenib (N=11)
rash/hand-foot syndrome (Skin and subcutaneous tissue disorders) | 6

LIMITATIONS AND CAVEATS:
The study was discontinued, after withdrawal from the sponsor due to slow accrual. The discovery of EGFR mutations changed the scope of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less